CLINICAL TRIAL: NCT03997435
Title: A Randomized Study of Neoadjuvant Chemoradiotherapy With or Without Intensification With the FOLFOXIRI Chemo-regimen for High-risk Locally Advanced Rectal Cancer
Brief Title: FOLFOXIRI With or Without Intensification for Rectal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: CCTU (Other)
Responsible Party: Sponsor-Investigator, CCTU, Comprehensive Cancer Trials Unit, Department of Clinical Oncology, The Chinese University of Hong Kong, Chinese University of Hong Kong
Organization: Chinese University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COL026
Record Dates: First submitted 2019-06-19; First posted 2019-06-25 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Rectal Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control arm (Experimental): neoadjuvant concurrent capecitabine-radiotherapy followed by surgery and postoperative chemotherapy
  Interventions: Drug: Control arm
- Experimental arm (Experimental): Neoadjuvant FOLFOXIRI x4 cycles, then capecitabine-radiotherapy and postoperative chemotherapy
  Interventions: Drug: Experimental arm

INTERVENTIONS:
Drug: Control arm — neoadjuvant concurrent capecitabine-radiotherapy followed by surgery and postoperative chemotherapy.
  Arms: Control arm
Drug: Experimental arm — Neoadjuvant FOLFOXIRI x4 cycles, then capecitabine-radiotherapy and postoperative chemotherapy.
  Arms: Experimental arm

SUMMARY:
Pathologic complete response rate

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent
* Age >= 18 years of either sex.
* ECOG performance status 0-1
* Measurable disease by RECIST 1.1 criteria.
* Histologically confirmed rectal adenocarcinoma (defined as either mid- or low rectal cancer that is located within 12 cm from the anal verge OR below the peritoneal reflection) that is previously untreated.
* 'High risk' rectal cancer, or rectal cancers that are considered marginally perable where there is a significant risk of positive surgical margin:
* T3 or T4, and / or
* Tumour infiltrating perirectal fat and/ or mesorectal fascia, and / or Involvement of pelvic lymph nodes, and/or
* Tumour invading surrounding structures or peritoneum or vasculature.
* Adequate bone marrow, renal and hepatic function as defined by: absolute neutrophil count >= 1.5 x 109/L, hemoglobin >= 9 g/L, platelets >= 100 x 109/L, serum creatinine level < 1.5 x ULN (or calculated creatinine clearance >=50 ml/min, whichever is worse), total bilirubin <=1.5 x the upper limit of normal, alanine aminotransferase (ALT) < 3 upper limit of normal.

Exclusion Criteria:

* Known distant metastasis, even if the metastasis has been resected.
* History of another invasive malignancy within the last 5 years, except for treated basal cell carcinoma of the skin, cervical intraepithelial neoplasia, or breast DCIS.
* Upper rectal cancer that is located above the peritoneal reflection.
* Patients with synchronous colon and rectal cancers are not excluded as long as: (1) these tumors are considered as two separate primaries (i.e. not metastasis or a contiguous part of a large primary), (2) both tumors are not causing imminent obstruction; (3) pelvic radiotherapy is not considered a contraindication.
* Primary tumour associated with any one of the following features:Frank intestinal obstruction, or
* Endoscope unable to pass through the tumour's lumen plus worsening local obstructive symptoms. Note: Patients with such features should be assessed by the surgical team regarding stomal bypass prior to study enrolment. Such patients can still be considered for study enrolment after undergoing stomal bypass.
* Known hypersensitivity reaction to the study drugs (i.e. fluoropyrimidine, irinotecan, oxaliplatin)
* Known peripheral neuropathy of grade 2 or more in severity.\ -Patients who have received an experimental anticancer therapy within the last 28 days.
* Previous pelvic radiotherapy
* Previous oxaliplatin or irinotecan for the treatment of colon or rectal cancer.
* Patient with hip prosthesis
* Major surgery (i.e. requiring general anaesthetics) within the last 28 days. Exception: Any patient who underwent stomal bypass for obstructing primary tumour within the last 14 days are still eligible, as long as the patient has sufficiently recovered from the surgery at the investigator's discretion.
* Known cardiac disease that is symptomatic or poorly controlled, including cardiac failure, arrhythmia or ischemic heart disease.
* Myocardial infarction or cerebrovascular accident within the last 12 months.
* Intercurrent infections or medical illnesses that are serious/ potentially life-threatening and require ongoing treatment.
* Patients who are unable to take capecitabine tablets uncrushed by the oral route (e.g. enteral feeding). Patients with significantly impaired gastrointestinal integrity and absorption are excluded.
* Patients with known and untreated bilateral hydronephrosis and/or hydroureters (or unilateral hydronephrosis and/or hydroureters in any patient with a single kidney) are excluded. The obstruction should be treated with ureteric stent(s) or percutaneous nephrostomy(s) prior to study enrolment. Patients with unilateral hydronephrosis and/or hydroureters and adequate renal function (i.e. as stated in the eligibility criteria: serum creatinine level < 1.5 x ULN, or calculated creatinine clearance >=50 ml/min - whichever is worse) are not excluded.
* Patients on warfarin therapy. Patients on low molecular weight heparin are not excluded.
* Pregnant or lactating women.
* Patients with reproductive potential who are not willing to use barrier method of birth control.
* Patients who are unable to provide written informed consent, or to comply with study requirements as judged by the investigator.
* Patients who refuse surgical treatment of the rectal cancer.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2019-09-10 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of pathologic complete response | 2 years

SECONDARY OUTCOMES:
Rate of tumour regression grade | 2 years
Number of objective tumour response | 2 years
Rate of circumferential resection margin (CRM) clearance | 2 years
Rate of tumour downstaging | 2 years
Number of Participants with Adverse Events | 2 years
Rate of overall survival | 5 years
Rate of disease-free survival, relapse-free survival | 5 years
Time to local (and distant) recurrence | 5 years
Number of patients with 30-days post-operative mortality | 1 month
Rate of compliance to study treatment | 2 years
Number of response to neoadjuvant therapy | 2 years

CONTACTS AND LOCATIONS:
Locations (3):
- Hong Kong (3):
  - Department of Clinical Oncology, Queen Mary Hospital, Hong Kong
  - Department of Oncology, Princess Margaret Hospital, Hong Kong
  - The Chinese University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No